CLINICAL TRIAL: NCT07272655
Title: A Prospective, Randomized, Double-Blind, Non-Inferiority Trial Comparing Ascending Aorta/Hemiarch Replacement Versus Total Arch Replacement With Frozen Elephant Trunk in Patients With Type A Aortic Intramural Hematoma
Brief Title: Hemiarch vs. Total Arch With FET for Type A Aortic IMH
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Hospital of Jilin University (Other)
Responsible Party: Principal Investigator, Kexiang Liu, MD, Department of Cardiovascular Surgery, Second Hospital of Jilin University, Second Hospital of Jilin University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: JDEYXWK305
Record Dates: First submitted 2025-11-26; First posted 2025-12-09 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-11

CONDITIONS: Type a Aortic Dissection
Keywords: Aortic Intramural Hematoma, Type A; Hemiarch Replacement; Total Arch Replacement; Non-Inferiority Trial; False Lumen Patency
MeSH Terms: conditions — Aortic Intramural Hematoma

STUDY DESIGN:
Intervention Model Description: This is a randomized, double-blind, parallel-group, non-inferiority trial. Participants are assigned 1:1 to receive either Ascending Aorta with Hemiarch Replacement or Ascending Aorta with Total Arch and Frozen Elephant Trunk Replacement.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participant Blinding: The patient will not be informed of whether they received a hemiarch or total arch replacement procedure. This is maintained through consistent post-operative communication that does not disclose the specific surgical technique.
  Outcome Assessor Blinding: The members of the independent imaging core laboratory, who are responsible for evaluating the primary endpoint (post-operative CTA scans for false lumen patency), are blinded to the patient's group assignment. All identifying information and surgical details related to the group allocation are removed from the images before analysis.
  Care Provider (Surgeon) Blinding: The operating surgeons cannot be blinded due to the nature of the surgical interventions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ascending Aorta / Hemiarch Replacement Group (Experimental): Participants randomized to this group will undergo Ascending Aorta and hemiarch replacement surgery. The procedure involves replacing the ascending aorta and the proximal portion of the aortic arch , while preserving the distal arch and supra-aortic vessels.
  Interventions: Procedure: Ascending Aorta / Hemiarch Replacement
- Total Arch Replacement and Frozen Elephant Trunk Replacement Group (Active Comparator): Participants randomized to this group will undergo conventional aortic total arch replacement surgery. This typically involves replacing the entire aortic arch , often combined with a frozen elephant trunk procedure into the descending aorta.
  Interventions: Procedure: Total Arch Replacement and Frozen Elephant Trunk Replacement.

INTERVENTIONS:
Procedure: Ascending Aorta / Hemiarch Replacement — This procedure involves the replacement of the ascending aorta and the proximal portion of the aortic arch (hemiarch). The distal aortic arch and the origins of the supra-aortic vessels (brachiocephalic trunk, left common carotid artery, and left subclavian artery) are preserved. It does not involve the implantation of a stent graft into the descending aorta.
  Other Names: Partial Arch Replacement
  Arms: Ascending Aorta / Hemiarch Replacement Group
Procedure: Total Arch Replacement and Frozen Elephant Trunk Replacement. — This procedure involves the replacement of the entire aortic arch, combined with the implantation of a frozen elephant trunk (FET) stent graft into the proximal descending aorta. The arch vessels are typically re-implanted as a single branch island patch or individually. The procedure includes total resection of the arch and aims to promote false lumen thrombosis in the proximal descending aorta.
  Other Names: Total Arch Replacement with FET
  Arms: Total Arch Replacement and Frozen Elephant Trunk Replacement Group

SUMMARY:
This is a prospective, randomized, double-blind, non-inferiority clinical trial designed to compare the efficacy and safety of two surgical strategies for Type A aortic intramural hematoma (TAIMH): (1) Ascending aorta /hemiarch replacement (A/HAR), and (2) Ascending aorta with total arch replacement and frozen elephant trunk (TARFET).

Patients with acute TAIMH will be enrolled based on computed tomography angiography (CTA) confirmation of a completely thrombosed false lumen in the ascending aorta and aortic arch. Eligible participants will be randomly assigned in a 1:1 ratio to either the A/HAR group (experimental) or the TARFET group (active comparator).

The primary endpoint is the rate of perioperative false lumen patency in the aortic arch and descending aorta, assessed postoperatively by a blinded, independent imaging core laboratory using CTA. Secondary endpoints include the aortic cross-clamp time, circulatory arrest time, total operation time, aortic reintervention rate, and perioperative complications, rate of false lumen patency in the aortic arch and descending aorta at 6 - 12 months.

The study tests the non-inferiority hypothesis that the less extensive A/HAR strategy is not inferior to the more extensive TARFET strategy in preventing early false lumen patency, while also exploring its potential superiority regarding other operative outcomes, such as reduced procedure times and lower incidence of complications. A total of 300 participants will be enrolled to ensure adequate statistical power. The findings from this trial are expected to provide high-quality evidence to guide optimal surgical strategies for patients with this unique aortic pathology.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years and ≤ 80 years.
2. Diagnosis of type A aortic intramural hematoma (TAIMH).
3. Ability to understand the study procedure and provide written informed consent.

Exclusion Criteria:

1. Preoperative CTA shows an open or partially thrombosed (mixed) false lumen in the ascending aorta or arch.
2. Primary tear located on the greater curvature of the aortic arch, necessitating total arch replacement.
3. Planned concomitant major cardiac surgery (e.g., CABG, valve replacement, atrial fibrillation ablation).
4. Previous history of aortic arch or distal aortic surgery.
5. Severe peripheral vascular disease or cerebrovascular anatomy abnormality.
6. Active systemic infection, malignancy, severe hepatic or renal dysfunction, or other major comorbidities with life expectancy < 1 year or deemed unfit for complex cardiovascular surgery.
7. Pregnancy or lactation.
8. Severe psychiatric or cognitive disorders affecting compliance or follow-up.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2027-04-20 (Estimated); Study Completion 2027-10-20 (Estimated)

PRIMARY OUTCOMES:
Rate of Perioperative False Lumen Patency in the Aortic Arch and Descending Aorta | At hospital discharge, an average of 5 to 14 days post-operatively
  This outcome measures the proportion of patients with patency (re-canalization) of the false lumen in both the aortic arch and descending aorta during the immediate postoperative period before hospital discharge.

SECONDARY OUTCOMES:
Aortic Cross-Clamp Time | Intraoperative period.
  Duration (minutes) of aortic cross-clamping during surgery.
Circulatory Arrest Time | Intraoperative period.
  Duration (minutes) of total circulatory arrest.
Total Operation Time | Intraoperative period.
  Total time (minutes) from skin incision to closure
Rate of Re-intervention on the Aorta | 6 months post-operatively
  The proportion of patients requiring any secondary surgical or endovascular procedure (e.g., TEVAR, open repair) specifically related to the aorta after the initial surgery
Perioperative Complications | 30 days after surgery
  incidence of major complications within 30 days post-surgery, including but not limited to neurological events, renal dysfunction, infection, bleeding, and cardiac failure.
rate of false lumen patency in the aortic arch and descending aorta at 6 - 12 months | One assessment performed between 6 and 12 months post-operatively.
  The proportion of patients with patency of the false lumen in the aortic arch and descending aorta, assessed at a single time point between 6 and 12 months after surgery during the follow-up period.

CONTACTS AND LOCATIONS:
Overall Officials: kexiang Liu, Ph.D., Principal Investigator — Department of Cardiovascular Surgery, The Second Hospital of Jilin University

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) that underlie the results reported in the published article will be shared. This includes baseline demographic data, clinical characteristics, operative details, and all primary and secondary outcome measures collected during the study. Additionally, the study protocol, statistical analysis plan (SAP), and clinical study report (CSR) will be made available to provide context for the data.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Beginning 6 months after the publication of the primary results and for a period of 5 years.
Access Criteria: Researchers with a methodologically sound proposal, approved by an independent review committee. Data requestors will be required to sign a data access agreement.